CLINICAL TRIAL: NCT05003102
Title: Dexmedetomidine Cycling and Sleep in the Pediatric ICU
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No enrollment, IRB closed
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Chiara Foster, MD, Pediatric Critical Care Medicine Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 210478
Record Dates: First submitted 2021-07-29; First posted 2021-08-12 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Critical Illness; Sedation Complication; Delirium
Keywords: dexmedetomidine; sleep
MeSH Terms: conditions — Critical Illness; Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: randomized crossover trial
Who Masked: Outcomes Assessor
Masking Description: Sleep study interpreters will not know which night had dexmedetomidine preferentially increased
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine cycling then Standard Pediatric Intensive Care Unit (PICU) sedation protocol (Experimental): One the first night, participants receive a dexmedetomidine bolus of 0.5 mcg/kg which is then titrated at an increased drip rate of 0.3 mcg/kg/hr until a.) a targeted Richmond Agitation-Sedation Scale (RASS) state that is one level deeper than what was targeted during the day is achieved or b.) infusion is at max drip rate (dexmedetomidine 2 mcg/kg/hr). On the second night, participants receive the standard PICU Sedation Protocol of fentanyl infusion at 1 mcg/kg/hr and dexmedetomidine infusion at 0.3 mcg/kg/hr with no modifications made until goal RASS reached or at max infusion drips achieved (fentanyl 5 mcg/kg/hr and dexmedetomidine 2 mcg/kg/hr).
  Interventions: Drug: Dexmedetomidine Hydrochloride - Cycling; Drug: Fentanyl - PICU Standard; Drug: Dexmedetomidine Hydrochloride - PICU Standard
- Standard Pediatric Intensive Care Unit (PICU) sedation protocol then Dexmedetomidine cycling (Active Comparator): On the first night, participants will receive the standard PICU Sedation Protocol of fentanyl infusion at 1 mcg/kg/hr and dexmedetomidine infusion at 0.3 mcg/kg/hr with no modifications made until goal RASS reached or at max infusion drips achieved (fentanyl 5 mcg/kg/hr and dexmedetomidine 2 mcg/kg/hr). On the second night, participants receive a dexmedetomidine bolus of 0.5 mcg/kg which is then titrated at an increased drip rate of 0.3 mcg/kg/hr until a.) a targeted Richmond Agitation-Sedation Scale (RASS) state that is one level deeper than what was targeted during the day is achieved or b.) infusion is at max drip rate (dexmedetomidine 2 mcg/kg/hr).
  Interventions: Drug: Dexmedetomidine Hydrochloride - Cycling; Drug: Fentanyl - PICU Standard; Drug: Dexmedetomidine Hydrochloride - PICU Standard

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride - Cycling — Dexmedetomidine Hydrochloride infusion at 0.5 mcg/kg titrated to 0.3 mcg/kg/hr up to a max drip rate of 2 mcg/kg/hr.
  Other Names: Precedex
Drug: Fentanyl - PICU Standard — fentanyl infusion at 1 mcg/kg/hr up to a max drip rate of 5 mcg/kg/hr
Drug: Dexmedetomidine Hydrochloride - PICU Standard — Dexmedetomidine Hydrochloride infusion at 0.3 mcg/kg titrated to 0.5 mcg/kg/hr up to a max drip rate of 2 mcg/kg/hr
  Other Names: Precedex

SUMMARY:
This is a study of mechanically ventilated pediatric intensive care unit (ICU) teenage patients and the effects of the medication dexmedetomidine on sleep, delirium, and sedation level. The Investigators will assess sleep with an 8 lead polysomnogram study and increase the medication at night for one night to see if the sleep architecture changes. The Investigators will assess their sleep with our unit's sedation protocol for an additional night.

DETAILED DESCRIPTION:
Background: Sleep deprivation is a common problem in the intensive care unit (ICU). Poor sleep is both a modifiable risk factor for improved recovery from severe illness and for delirium which is associated with increased mortality (1, 2). Sleep deprivation is a physiological stressor that can affect the autonomic, immune, metabolic, and hormonal functions of the body. Inflammatory cytokines are increased during sleep deprivation and hormonal responses to stress which are already affected by critical illness are worsened with lack of sleep (3, 4).

Sedation greatly confounds the ability to distinguish if a patient is asleep or simply deeply sedated particularly in the mechanically ventilated pediatric population. Kudchadkar et.al looked at sleep architecture using limited montage electroencephalogram and saw that sleep was abnormal on sedative infusions although this study did not look at dexmedetomidine infusion (5). However, polysomnography as the gold standard to asses sleep can offer more details about sleep architecture including arousal index. It is well known that sedatives have natural sleep properties, but The Investigators do not have much data on how they impact sleep architecture in the pediatric population. When attempting to describe sleep in the ICU, sleep is inaccurately determined by bedside providers clinically (6-8). The age and severity of illness of intubated pediatric patients them poor candidates for self-reporting using a behavioral scales to describe sleep. Evaluating sleep using polysomnography both removes observer inaccuracy and provides information on the sleep architecture of patients on sedative infusions.

Dexmedetomidine is a commonly used infusion for sedation in the ICU that also has natural sleep properties. It is an alpha 2 agonist that acts at the locus coeruleus which is involved in arousal (9). It mimics natural sleep in animal models (10). Dexmedetomidine is commonly used in pediatric intensive care units, although its use has gained increased popularity in the last five years. While some pediatric intensivists cycle, increase the dose at night, of dexmedetomidine to reduce delirium, there is only adult data describing an association between nocturnal dexmedetomidine infusion and reduced delirium (11,12). There are no studies published assessing sleep architecture via polysomnography in pediatric patients on dexmedetomidine infusions. The Investigators aim to assess sleep architecture as well as incidence of delirium in patients who have dexmedetomidine infusions increased during nocturnal hours.

It is well established that critically ill children and adults have poor sleep quality and quantity during an ICU stay. Emerging research suggests sleep may improve patient outcomes by mitigating negative effects of the ICU environment such as delirium. Many of the sedatives used in the ICU may disrupt sleep architecture, but pharmacologic studies suggest the sedative dexmedetomidine may improve sleep. Clinical studies in critically ill adults have shown benefit to using dexmedetomidine sedation overnight, or by increasing the dose at night for patients receiving continuously. Pediatric intensivists have started increasing dexmedetomidine infusion doses at night for delirious patients with anecdotal improvements in mental status and delirium state the following day, but no evidence has been published to support this practice.

Study: The purpose of this small pilot study is to assess if nocturnal sleep quality and quantity improves with increasing the dose of continuous intravenous infusion of dexmedetomidine exclusively to attain a targeted Richmond Agitation Sedation Scale (RASS) state in intubated and critically ill pediatric patients between the age of 12 and 17 in the pediatric intensive care unit instead of utilizing increasing doses of 2-3 agents with dexmedetomidine being one of them. The FDA has not approved this medication for use in children, so this study will only enroll patients already placed on the medication by their care team as it is already used by this unit in spite of lack of FDA approval for pediatrics. An Investigational New Drug (IND) application was submitted to the FDA and this study was deemed IND exempt (IND 155894). For the control night, the Investigators will make no modifications to the Vanderbilt Children's Hospital approved pediatric intensive care unit sedation protocol. The Investigators will use the same titration and approved maximum doses which are as follows: Initiate fentanyl infusion at 1 mcg/kg/hr and dexmedetomidine infusion at 0.3 mcg/kg/hr, if RASS greater than desired RASS implement the following in order until RASS goal is met. Step 1: Give fentanyl bolus of 1 mcg/kg, reassess in 10 minutes; Step 2: Repeat fentanyl bolus of 1 mcg/kg and increase drip by 1 mcg/kg/hr, reassess in 10 minutes; Step 3: Give dexmedetomidine bolus of 0.5 mcg/kg, reassess in 10 minutes; Step 4: Repeat dexmedetomidine bolus of 0.5 mcg/kg and increase drip by 0.3 mcg/kg/hr, reassess in 10 minutes. Repeat steps 1-4 until goal RASS reached or at max drips (fentanyl 5 mcg/kg/hr and dexmedetomidine 2 mcg/kg/hr). For the intervention night, the Investigators will use the same titration and maximum dose of dexmedetomidine that is Vanderbilt Children's Hospital approved. The Investigators will start the dexmedetomidine where the patients daytime providers have dosed it and titrate to a targeted RASS goal one level deeper. The Investigators will follow the unit titration of using 0.5 mcg/kg bolus and increasing the drip by 0.3 mcg/kg/hr. Reassess RASS 10 minutes later, and if not at desired RASS goal, repeat bolus of 0.5 mcg/kg and increase by 0.3 mcg/kg/hr until either the desired RASS goal is met or a maximum of 2 mcg/kg/hr is reached.

The Investigators aim to enroll children who are currently receiving mechanical ventilation and dexmedetomidine infusion for sedation per current pediatric ICU practice and assess the effects of preferentially increasing dexmedetomidine infusion on nocturnal sleep architecture. The Investigators will assess sleep using an 8 lead montage of polysomnography. Each patient will wear the polysomnogram leads for two nights. One of the two nights will follow the intensive care unit sedation protocol (allowing for use of other sedatives as needed) versus increasing the dose of dexmedetomidine to a target Richmond Agitation-Sedation Scale state one level deeper than what was targeted during the day. Those interpreting the sleep studies will be blinded to which night was the night that the dexmedetomidine infusion was preferentially increased.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are intubated and ages 12 years and 0 days old to 17 years and 364 days old who are admitted to the Pediatric intensive care unit and who are on the sedation protocol with use of at least an intravenous dexmedetomidine infusion
* Patients will be selected from those admitted from the emergency room for traumas and critical illness as well as those admitted for post-operative care
* Prematurity, history of permanent neurological damage, autism spectrum disorder, presence of genetic conditions will not preclude enrollment

Exclusion Criteria:

* Patients taking clonidine daily prior to admission
* Those with allergy to dexmedetomidine
* Those on non-intravenous forms of dexmedetomidine
* Those on a ketamine, propofol, pentobarbital, or paralytic infusions
* Those with a diagnosis of refractory status epilepticus
* Patients with vision loss
* Those admitted for care following a cardiac arrest
* Those with a history of hemodynamic instability with dexmedetomidine infusion and lack of a permanent pacemaker or implantable cardioverter-defibrillator
* Those with International Normalized Ratio (INR) >3.2 (due to concerns for reduction in clearance by 50% in pediatric patients at that level of coagulopathy)
* Those on antiarrhythmics (due to association with cardiac arrest with dexmedetomidine and amiodarone and concerns with administration while on digoxin)
* Those with a Glascow Coma Scale (GCS) of 3T or less at presentation
* Those on sedation for end of life comfort

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in total sleep time as seen via an 8-lead polysomnogram | 2200 hours to 0600 hours during each study night; up to 2 study nights during the hospital admission
  quantitative measure of physiological parameter; sleep software will add all sleep time together for final value in hours and minutes
Change in total time in different stages of sleep as seen via an 8-lead polysomnogram | 2200 hours to 0600 hours during each study night; up to 2 study nights during the hospital admission
  quantitative measure of physiological parameter; sleep study interpreter will determine time spent in stages N1, N2, N3, and Rapid Eye Movement (REM) based upon architecture of the sleep spindles and add together for final amount of time in hours and minutes spent in each stage
Change in arousal index as seen via an 8-lead polysomnogram | 2200 hours to 0600 hours during each study night; up to 2 study nights during the hospital admission
  quantitative measure of physiological parameter; sleep study interpreter will determine the number of arousals and awakenings and divide this by the total sleep time

SECONDARY OUTCOMES:
Incidence of Delirium | Day 1 between 0800 hours and 1900 hours; Day 1 between 1900 hours and 0800 hours; and Day 2 between 0800 hours and 1900
  nurse completes the 2 step, 4 feature, 5 question Pediatric (or the 2 step, 4 feature, 6 question preschool if patient has developmental delays that place patient at a preschool level) Confusion Assessment Method for the Intensive Care Unit on patient. Step 1 looks at if the patient is arousable and if so then the screener goes to step 2 with the 4 features of 'yes or no' questions. Feature 1 has 2 questions about change or fluctuation in mental status baseline. If both are no, patient is scored as "delirium absent" and screening is complete. If yes, the 3 other features are performed which look at inattention, altered level of consciousness, and disorganized brain. The nurse assesses the patients ability to complete tasks in features 2 and 4 in the pediatric version and in feature 2 in the preschool version. If the answer is yes in the features, patient scores as "delirium present".
Sedation Exposure | 2200 hours to 0600 hours each study night; up to 2 study nights during the hospital admission
  quantitative measure; will review medication administration record and count the number of recorded boluses of sedation medications given that night

CONTACTS AND LOCATIONS:
Overall Officials: Chiara N Foster, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers

REFERENCES:
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Figueroa-Ramos MI, Arroyo-Novoa CM, Lee KA, Padilla G, Puntillo KA. Sleep and delirium in ICU patients: a review of mechanisms and manifestations. Intensive Care Med. 2009 May;35(5):781-95. doi: 10.1007/s00134-009-1397-4. Epub 2009 Jan 23. PMID 19165463
- [Background] Faraut B, Boudjeltia KZ, Vanhamme L, Kerkhofs M. Immune, inflammatory and cardiovascular consequences of sleep restriction and recovery. Sleep Med Rev. 2012 Apr;16(2):137-49. doi: 10.1016/j.smrv.2011.05.001. Epub 2011 Aug 10. PMID 21835655
- [Background] Vgontzas AN, Zoumakis E, Bixler EO, Lin HM, Follett H, Kales A, Chrousos GP. Adverse effects of modest sleep restriction on sleepiness, performance, and inflammatory cytokines. J Clin Endocrinol Metab. 2004 May;89(5):2119-26. doi: 10.1210/jc.2003-031562. PMID 15126529
- [Background] Kudchadkar SR, Yaster M, Punjabi AN, Quan SF, Goodwin JL, Easley RB, Punjabi NM. Temporal Characteristics of the Sleep EEG Power Spectrum in Critically Ill Children. J Clin Sleep Med. 2015 Dec 15;11(12):1449-54. doi: 10.5664/jcsm.5286. PMID 26194730
- [Background] Kamdar BB, Shah PA, King LM, Kho ME, Zhou X, Colantuoni E, Collop NA, Needham DM. Patient-nurse interrater reliability and agreement of the Richards-Campbell sleep questionnaire. Am J Crit Care. 2012 Jul;21(4):261-9. doi: 10.4037/ajcc2012111. PMID 22751369
- [Background] Hoey LM, Fulbrook P, Douglas JA. Sleep assessment of hospitalised patients: a literature review. Int J Nurs Stud. 2014 Sep;51(9):1281-8. doi: 10.1016/j.ijnurstu.2014.02.001. Epub 2014 Feb 15. PMID 24636444
- [Background] Richardson A, Crow W, Coghill E, Turnock C. A comparison of sleep assessment tools by nurses and patients in critical care. J Clin Nurs. 2007 Sep;16(9):1660-8. doi: 10.1111/j.1365-2702.2005.01546.x. Epub 2007 Apr 24. PMID 17459137
- [Background] Weerink MAS, Struys MMRF, Hannivoort LN, Barends CRM, Absalom AR, Colin P. Clinical Pharmacokinetics and Pharmacodynamics of Dexmedetomidine. Clin Pharmacokinet. 2017 Aug;56(8):893-913. doi: 10.1007/s40262-017-0507-7. PMID 28105598
- [Background] Nelson LE, Lu J, Guo T, Saper CB, Franks NP, Maze M. The alpha2-adrenoceptor agonist dexmedetomidine converges on an endogenous sleep-promoting pathway to exert its sedative effects. Anesthesiology. 2003 Feb;98(2):428-36. doi: 10.1097/00000542-200302000-00024. PMID 12552203
- [Background] Skrobik Y, Duprey MS, Hill NS, Devlin JW. Low-Dose Nocturnal Dexmedetomidine Prevents ICU Delirium. A Randomized, Placebo-controlled Trial. Am J Respir Crit Care Med. 2018 May 1;197(9):1147-1156. doi: 10.1164/rccm.201710-1995OC. PMID 29498534
- [Background] Hong KS, Kim NR, Song SH, Hong G. Cycling of Dexmedetomidine May Prevent Delirium After Liver Transplantation. Transplant Proc. 2018 May;50(4):1080-1082. doi: 10.1016/j.transproceed.2017.11.076. PMID 29731070
- See also: FDA Sheet for Dexmedetomidine Hydrochloride (Reference ID: 3836249) — https://www.accessdata.fda.gov/drugsatfda_docs/label/2015/206628s000lbl.pdf